CLINICAL TRIAL: NCT05298865
Title: Addressing Stress-induced Decision-making Bias in Parents for Promoting COVID-19 Vaccination Among Hong Kong Children: a Survey-based Experiment
Brief Title: Parental Health Decision-making for Children During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 20220113pavdm
Record Dates: First submitted 2022-03-23; First posted 2022-03-28 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Stress; Coping Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutral recall message (Placebo Comparator): Control group will receive a set of messages guiding them to recall neutral life senarios/objects. The messages will contain eight brief paragraphs of neutral text and icon-based pictures to guide participants to recall their life senarios. The text message will include yesterday's meals, yesterday's wearing, home environment and nearby locations. This control condition equated attention and time on task but expect not to induce any emotions in participants.
  Interventions: Behavioral: Neutral recall message
- Positive imagination stimulation (Experimental): Positive-affect-priming group (PA) will receive a set of messages guiding participants to imagine positive future life senarios. Prior receiving the PA messages, a brief instruction will also be provided to guide participants to imagine concrete and personal images while browsing the following messages. The PA messages will contain eight pictures representing the life senarios and accompanying with short text to guide participants' imagination. Each senario will contain two pictures, one is used to familiarized participants with the context that they are going to imagine (i.e. imagine one of your best friends); the second one provides richer information to stimulate participants' concrete imagination (i.e. imagine you share a good news with your friend). These intervention messsages aim to intentionally manipulate participants' feelings arousal and mental representation for positive future life.
  Interventions: Behavioral: Positive imagination stimulation

INTERVENTIONS:
Behavioral: Positive imagination stimulation — The intervention messages aim to generate participants' positive mental image toward their life and also to relieve parental stress by shifting their attention to positive life events. The positive affect cues will be developed based on qualitative interviews with 30 parents from our previous study during pandemic and also extended literatures on positive psychology. Our previous qualitative interview aimed to understand parental concerns on flu and COVID-19 vaccination, parental life stressors throughout the pandemic were also explored. The positive cues will be discussed and evaluated by the research team with an aim to cover major positive life events that are personal relevant to parents, including positive social support (friendship), positive family support (family gathering), qualified time spent with children (here we will also embed a gratitude practice to elicit strong positive feelings), and cultivate positive self by imagining achieving personal goals in the future.
  Arms: Positive imagination stimulation
Behavioral: Neutral recall message — The control message aims to equate time and attention as in the intervention group. Therefore, a recall task will be assigned to participants. Brief texts will be provided to guide participants to memorize their life senarios but not to induce emotions. Messages include the following: recall the breakfast and lunch you had yesterday; recall the clothes and shoes you wore yesterday; recall the kitchen in your home; recall one of the chairs in your home; recall the routes to the nearest supermarket and subway of your house.
  Arms: Neutral recall message

SUMMARY:
Background: As major decision-maker for children's wellbeing, parents play a vital role in decisiding on a wide range of health-related issues including vaccination. Such decision-making process will be complicated by a great amount of psychosocial stressors emerging from the current pandemic. Stress can lead to various decision-making biases for children vaccination and subsequently lead to low vaccination intention amongst parents, which may hinder the progress for reaching herd immunity and end the COVID-19 pandemic. Effective risk communication intervention thus is in urgent need to address stress-induced decision-making biases for an upcoming COVID-19 vaccine for young children.

Aims: This study will investigate the interrelationships among parental perceived stress, and interpretive bias toward negative vaccine-related stimuli and and vaccination intention. In addition, this study will also conduct a survey experiment to develop positive affect-based messages and test its effect on correcting stress-induced biases in vaccination decision making among parents with high mental stress level.

Design and subjects: We aim to recruit parents aged 18 years or above with at least one child in our study. Participants will be recruited from our previous study through WhatsApp. Participants will be invited to read a list of vaccine-related news headlines with a mixture of positive and negative sentiments first. Then they will be asked to complete a series of assessment on their vaccination decision-making and intention. In the next phase, a survey-based experiment will be embedded in the online questionnaire to test the effect of risk communication interventions. Intervention messages will be designed based on previous qualitative study and literatures on positive psychology to simulate parents' positive mental images of COVID-19 vaccination consequences by using positive-affect visual stimuli.

Main outcome measures and analysis: Participants will be invited to complete a series of assessments through online questionnaire to assess their mental stress level, negative interpretive bias on processing ambiguous vaccine information and behavioural intention for vaccinating children.

Paired t-test will be used to determine negative interpretive bias between high-stress vs. low-stress parents. Structural equation modelling (SEM) will be performed to test the relationships among parental mental stress level, affect-driven decision-making constructs and vaccination intention for children. For the survey-based experiment, the effect of positive-affect messages intervention on tendency of correcting decision-making biases and COVID-19 vaccine uptake for children will be evaluated using logistic regression model with perceived stress level and intervention as the main between-group factors.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one child aged below 12 years old;
* Hong Kong resident；
* Able to communicate in Cantonese, Mandarin or English;
* Capable of completing online questionnaire via WhatsApp.

Exclusion Criteria:

* Subjects with cognitive and linguistic difficulties prohibiting completing the interview will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Negative interpretive bias | Immediately after they complete the task with priming manipulation
  The negativity processing bias will be assessed by participants' subjective rating on a set of ambiguous news regarding the current pandemic. All the news will be adapted from real local news to simulate a natural news environment for participants. All the news will contain two parts, the former part will be risk-focused (more negative) while the latter part will be solution-focused (more positive). After reading 3 pieces of news, participants will be asked to rate how positive or negative of the news and how they feel about the news (valence and affective respond will be rated on a 7-point slider, -3 indicates very negative/pessimistic; 0 indicates neutral; 3 indicates very positive/optimistic). An additional question will be asked to assess participants' perceived self-efficacy after reading the news (scale 1-5, 1 indicates No confidence at all; 5 indicates Very confident). The valence, affect and self-efficacy scores for the 3 news will be summed into a single index for analysis

SECONDARY OUTCOMES:
Parental vaccine-hesitant attitudes after two weeks. | Two weeks after priming manipulation
  The parental vaccine-hesitant attitudes will be assessed using a 5-point Likert scale (1-5). Five statements are shown and the participants will be asked to rate the degree to which they agree or disagree with the statements. With 1 indicating Strongly disagree and 5 indicating Strongly agree.
Parental Mental Health Status | Two weeks after priming manipulation
  The parental mental health status will be assessed by Patient Health Questionnaire-4 (PHQ-4) two weeks after priming manipulation. The questionnaire contains 4 items describing different mental state (e.g. Feeling nervous, anxious or on edge) and the participants will be asked to rate how close these 4 items match their own situation in the past two weeks on a 4-point Likert scale (from 0-3). With 0 indicating Not at all and 3 indicating Nearly every day.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong School of Public Health, Hong Kong, Hong Kong